CLINICAL TRIAL: NCT02582931
Title: Pilot Study of MRI-Guided Stereotactic Body Radiation Therapy (SBRT) for Ovarian Cancer
Brief Title: MRI-Guided Stereotactic Body Radiation Therapy (SBRT) for Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201510101
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Cancer of Ovary; Cancer of the Ovary; Neoplasms, Ovarian; Ovarian Cancer; Ovary Cancer; Ovary Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Arm 1: MRI-guided SBRT (Experimental): * Radiotherapy will consist of stereotactic body therapy, to be given over five fractions, delivered once daily or once every other day for a period of one to two weeks, for a total of five treatments.
  * Patients will be planned for an initial dose of 35Gy to the planning target volume (PTV), with dose adaptation and reduction allowed based on safety constraints that are generally accepted, up to a maximum allowed total dose of 50Gy in five fractions to the PTV.
  * All patients will undergo both CT and MRI simulation in positioning appropriate for the specific treatment site
  Interventions: Device: MRI-guided SBRT; Behavioral: EORTC QLQ-C30 Questionnaire; Behavioral: EORTC QLQ-OV28 Questionnaire

INTERVENTIONS:
Device: MRI-guided SBRT
  Other Names: MRI-guided stereotactic body radiation therapy
Behavioral: EORTC QLQ-C30 Questionnaire — 30 questions with 28 questions having answers that range from 1 (not at all) to 4 (very much) and the other 2 questions have answers that range from 1 (very poor) to 7 (excellent)
Behavioral: EORTC QLQ-OV28 Questionnaire — 28 questions having answers that range from 1 (not at all) to 4 (very much)

SUMMARY:
The investigators propose to evaluate the feasibility, safety, and preliminary efficacy of delivering online, adaptive magnetic resonance imaging (MRI)-guided and gated stereotactic body radiation therapy for patients with recurrent or metastatic ovarian cancer on a novel, integrated Co-60 MRI treatment machine. To best assess this technology, the investigators will focus on patients that have no more than three sites of progressive disease within the central thorax, liver, and/or non-liver abdominopelvis to receive adaptive, MRI-guided and gated SBRT with MRI simulation. Patients will be treated in five fractions over one to two weeks. By adhering to strict normal tissue constraints, expected toxicity will be within the current standard of care but will allow adaptation based on daily anatomic changes. The prescription dose will be determined based on hard normal tissue constraints, and capped at 10Gy per fraction. Although the long term goal will be to achieve improved local control and disease-free survival with reduced toxicity, the present study will be driven by the short term goal of demonstrating the feasibility of this novel treatment approach for recurrent or metastatic ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed primary disease histology of solid ovarian, fallopian tube, or primary peritoneal tumor categorization.
* Deemed medically fit for stereotactic body radiation therapy by the treating physician.
* At least 18 years old.
* Karnofsky Performance Status ≥ 70
* Completed any systemic therapy (excluding endocrine therapy, which may be ongoing) at least one week prior to planned start of SBRT (two weeks preferred) and must have no plans to initiate systemic therapy for at least one week following end of SBRT (two weeks preferred).
* Able to understand and be willing to sign an IRB approved written informed consent document (or legally authorized representative, if applicable).

Exclusion Criteria:

* Past history of radiotherapy within the projected treatment field of any of the disease sites to be treated by MRI-guided, gated, and/or online adaptive SBRT
* Current central nervous systemic disease.
* Widespread progressive disease, i.e., more than three sites of progressive disease (note that more than three sites of disease are permitted provided there are no more than three sites of progressive disease).
* Actively receiving any investigational agents.
* Presence of uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Patients of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Medical contraindication to undergoing MR imaging.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of providing online, adaptive MRI-guided and gated SBRT as measured by the ability to deliver a full course of MRI-guided SBRT in at least 80% of eligible patients who have completed simulation and planning | Completion of all enrolled patients (up to 2 years)

SECONDARY OUTCOMES:
Safety as measured by acute toxicities | Up to 90 days post completion of treatment
  the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Safety as measured by late toxicities | 91 days to 6 months post completion of treatment
  the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Response rate | 3 months post treatment
  -Response will be measured using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009].
In-field control rate | 6 months post treatment
Local control rate | 3 months post treatment
Regional control rate | 3 months post treatment
Distant control rate | 3 months post treatment
Progression-free survival (PFS) rate | 6 months post treatment
  -PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Disease-free survival (DFS) rate | 6 months post treatment
  -The length of time that a patient survives without any signs or symptoms of their cancer
Overall survival (OS) rate | 6 months post treatment
Patient-reported health-related quality of life (HRQOL) | 6 months post treatment
  * HRQOL will be measured using the EORTC QLQ-C30 and QLQ-OV28 questionnaires.
  * European Organization for Research and Treatment of Cancer (EORTC) QLQ-30 consists of 28 questions with answers that range from 1 (Not At All) to 4 (Very Much) and 2 questions that range from 1 (Very Poor) to 7 (Excellent)
  * EORTC QLQ-OV28 consists of 28 questions ranging with answers from 1 (Not At All) to 4 (Very Much)
CA-125 response levels | 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Robinson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu